CLINICAL TRIAL: NCT03582007
Title: A Multicenter, Open Label, Sponsor Blinded, Randomized, Active Controlled, Parallel Group, Pivotal Study to Evaluate the Efficacy, Safety, and Tolerability of Murepavadin Given With Ertapenem Versus an Anti-pseudomonal-β-lactam-based Antibiotic in Adult Subjects With Nosocomial Pneumonia Suspected or Confirmed to be Due to Pseudomonas Aeruginosa
Brief Title: Pivotal Study in Nosocomial Pneumonia Suspected or Confirmed to be Due to Pseudomonas
Acronym: PRISM-UDR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety data review
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POL7080-010
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-05

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — murepavadin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Sponsor blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Murepavadin (Experimental): Murepavadin + ertapenem
  Interventions: Drug: Murepavadin
- Anti-pseudomonal antibiotic (Active Comparator): One anti-pseudomonal-β-lactam-based antibiotic (either meropenem or piperacillin-tazobactam)
  Interventions: Drug: One anti-pseudomonal antibiotic

INTERVENTIONS:
Drug: Murepavadin — Murepavadin + ertapenem
  Arms: Murepavadin
Drug: One anti-pseudomonal antibiotic — Either meropenem or piperacillin-tazobactam
  Arms: Anti-pseudomonal antibiotic

SUMMARY:
This is a phase 3, multicenter, open-label, sponsor blinded, randomized active-controlled, parallel group to investigate the efficacy, safety and tolerability of intravenous murepavadin given with ertapenem versus an anti-pseudomonal β-lactam based antibiotic in the treatment of nosocomial pneumonia in adult subjects

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has received mechanical ventilation for at least 48h at the time of the randomisation OR at least 2 of the following signs or symptoms presenting within 24 hours prior to randomization: New onset of cough or worsening of baseline cough and/or dyspnea, tachypnea and/or hypoxemia and/or new onset of sputum or suctioned respiratory secretion characterized by purulent appearance indicative of bacterial infection or a worsening in character of purulent appearance
* Acute Physiology and Chronic Health Evaluation (APACHE) of 8 to 25, inclusive, within 24h prior to randomization
* Presence of new or progressive infiltrate on chest X-ray
* Presence of clinical criteria consistent with Pneumonia
* Strong clinical suspicion of pneumonia due to P. aeruginosa

Key Exclusion Criteria:

* Known or suspected community-acquired bacterial pneumonia or viral, fungal, or parasitic pneumonia
* known hypersensitivity to any component of ertapenem, meropenem or to other drugs in the same class or demonstrated anaphylactic reactions to beta-lactams or a history of allergic reactions to any of the penicillins, cephalosporins, or β-lactamase inhibitors
* Severe liver or renal impairment
* Expected survival < 72 hours
* Evidence from an available surveillance culture of co infection with ertapenem , meropenem or piperacillin tazobactam resistant Gram negative pathogen(s)
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
All cause mortality rates | 28 days after start of study treatment

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - Research site, Iowa City, Iowa
  - Research Site, Pittsburgh, Pennsylvania
- Czechia (2):
  - Research site, Břeclav
  - Research site, Kolín
- Research site, Argenteuil, France
- Israel (2):
  - Research site, Hadera
  - Research site, Tel Aviv